CLINICAL TRIAL: NCT00882804
Title: Effect of Hemin on Heme-Oxygenase-1 Activity in Healthy Subjects
Brief Title: Hemin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Adil E. Bharucha, M.D., Mayo Clinic, Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 09-000230
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Healthy Volunteers
Keywords: hemin, heme oxygenase, humans, HO-1

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Hemin (Experimental)
  Interventions: Drug: Hemin infusion
- placebo (Placebo Comparator)
  Interventions: Drug: placebo infusion

INTERVENTIONS:
Drug: Hemin infusion — Hemin (Panhematin®, Ovation Pharmaceuticals, Deerfield, IL) will be administered through a large-caliber peripheral vein at a dose of 1.25 mL/kg and at a rate of 60 mL/hour. To enhance stability, Panhematin® will be diluted in ~ 132 mL of 25% albumin to obtain a hemin concentration of 2.4 mg/mL.
  Arms: Hemin
Drug: placebo infusion — 25 % albumin will be administered through a large-caliber peripheral vein at a dose at a rate of 60 mL/hour.
  Arms: placebo

SUMMARY:
This study is being done because we want to learn if hemin can increase the production of heme oxygenase 1. Heme oxygenase 1 (HO-1) is an enzyme which protects cells from physical, chemical, and biologic stress. Hemin is produced from red blood cells and is approved by the Food and Drug Administration for treating acute porphyria, which is an inherited condition caused by an enzyme deficiency.

DETAILED DESCRIPTION:
Heme-oxygenase 1 (HO-1) degrades heme, protects cells against oxidative stress, and is beneficial in several experimental models but has not been pharmacologically activated in humans. The objectives of this study were to evaluate the effects of hemin on HO-1 activity in healthy subjects. Hemin is the most powerful inducer of HO-1. Hemin is FDA-approved to treat acute intermittent porphyria. In addition, hemin has also been used to treat thalassemia intermedia, myelodysplastic syndrome, and to control liver allograft failure due to recurrence of erythropoietic prototheria. Our hypothesis is that compared to placebo, hemin will increase HO-1 in humans. Ten healthy subjects will be randomized to hemin (n = 5, Panhematin®, Ovation Pharmaceuticals, 3 mg/kg i.v. in 25% albumin) or placebo (n = 5, 25% albumin) infusion. HO-1 activity will be assessed before and after (4, 6, 24, and 48 hours) infusions.

ELIGIBILITY:
1. Healthy non pregnant not breast feeding, and non-smoking subjects aged 18 - 65 years old without clinical evidence of significant cardiovascular, gastrointestinal, hematological, neurological, psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns. No symptoms of functional GI disorder as assessed by a validated questionnaire.
2. No medications except for stable doses of oral contraceptives or thyroid supplementation. Because ascorbic acid can induce HO-1 activity, multivitamins will need to be discontinued for 1 week before and for the duration of the study.
3. No intolerance or allergy to eggs
4. Able to provide written informed consent before participating in the study
5. Able to communicate adequately with the investigator and to comply with the requirements for the entire study
6. Screening weight < 96 kg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Venous carboxyhemoglobin concentrations | at 6 hours
HO-1 protein concentration in leukocytes from venous blood | at 6 hours
Serum bilirubin | at 6 hours

SECONDARY OUTCOMES:
Venous carboxyhemoglobin concentrations | at 4, 24, and 48 hours
HO-1 activity in leukocytes from venous blood | at 4, 24, and 48 hours
Serum bilirubin | at 4, 24, and 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Adil E Bharucha, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States